CLINICAL TRIAL: NCT06743451
Title: Enhancing Growth Monitoring Visits Through Health Workers Training on Growth Monitoring and Promotion, GMP Guideline a Community Health Volunteer Mobilization for Increasing Demand of GMP Through GMP Day in Joshipur Rural Municipality, Kailai, Nepal
Brief Title: Enhancing Growth Monitoring Visits in Joshipur Rural Municipality, Kailai, Nepal
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kathmandu University School of Medical Sciences (Other)
Responsible Party: Principal Investigator, Amrita Ghimire, Lecturer (Public Health), Kathmandu University School of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: GMP2025
Record Dates: First submitted 2024-12-10; First posted 2024-12-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Malnourished Children
Keywords: Nepal; Growth monitoring and Promotion; Malnutrition
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Health workers of Joshipur rural municipality and Female community health volunteers (Experimental): Health workers will receive Training on GMP guideline, while FCHV will be mobilized for inviting mothers and caretakers having under two years children.
  Interventions: Other: Health workers training on GMP guideline; Other: Female community health volunteers' mobilization for inviting mothers and caretakers

INTERVENTIONS:
Other: Health workers training on GMP guideline — One day training will be conducted to health workers on updated GMP guideline for the health workers primarily engaged in Growth monitoring and promotion of the children.
Other: Female community health volunteers' mobilization for inviting mothers and caretakers — Female community health volunteers will be mobilized for inviting mothers and caretakers for two consecutive months for enhancing GMP practices in the municipality

SUMMARY:
The goal of this clinical trial is to learn if health workers training on growth promotion and monitoring guideline and Female Community Health Volunteers mobilization for increasing demand for growth monitoring and promotion, GMP through growth monitoring and promotion day, GMP day) can enhance the growth monitoring and promotion practices in mothers and caretaker having under two years children. The main questions it aims to answer are:

* Does health workers training on GMP guideline enhances the growth monitoring and promotion practices in mothers and caretakers having under two years children?
* Does FCHV mobilization enhances growth monitoring and promotion practices in mothers and caretakers having under two years children? Participants will
* Health workers of the Joshipur rural municipality will have to attend Training session on GMP guideline,
* Mothers and caretakers having under two years children will have to visit to the nearest health facility for GMP visits for their children

DETAILED DESCRIPTION:
For addressing the problem of malnutrition in the municipality, determinants of the problem have been identified through CFIR framework. Based on the identified facilitator and barriers, two strategies have been developed for solving the problem of the municipality- (a) health workers training on latest GMP guideline to update the knowledge and skills of the service providers (b) For increasing demand generation, inviting mothers and caretakers having under two years children

1. Health workers Training on GMP guideline: Mr. Ashish Timalsina will be responsible for one day training on GMP guideline to the health workers of all six health facilities who are primarily engaged in nutrition in Joshipur rural municipality.
2. FCHV mobilization for increasing demand of growth monitoring and promotion through GMP day: Particular days of the month will be specified as GMP day in the municipality. Mothers and caretakers having under two years children. Health coordinator of the Joshipur rural municipality will be responsible for monitoring and supervision of this strategy.

Objectives General Objective

● To assess the implementation outcomes of Health workers Training on GMP guidelines and FCHV mobilization for increasing demand of Growth monitoring and Promotion through GMP day.

Specific Objectives

* To assess acceptability, appropriateness, feasibility, fidelity of (a) Health workers Training on GMP guideline; and acceptability, appropriateness, feasibility of (b)FCHV mobilization for increasing demand of Growth monitoring and Promotion through GMP day by using PROCTOR's framework.
* To assess the effectiveness of interventions- Health workers Training on GMP guideline and FCHV mobilization for increasing demand of Growth monitoring and Promotion through GMP day by average number of GMP visits.

  6. Methodology

Study site and its justification:

The study site will be Joshipur rural municipality, Kailali. There are seven wards in Joshipur Rural Municipality, in which a total of six health facilities are providing services in the Municipality. Average growth monitoring visit of the municipality was only 8 visits per child out of 24 visits per child (who have completed two years) in the fiscal year 2079/80 BS (2022 AD). The practice of growth monitoring was only 43% in the fiscal year 2079/80 BS (2022 AD). (HMIS)

ELIGIBILITY:
Inclusion Criteria:

For Health Workers:

1. Nutrition focal person of the health facility having primary engagement in growth monitoring and promotion.
2. Trained on growth monitoring and promotion guideline.

For Female Community Health Volunteers 1. Active for inviting mothers and caretakers of the municipality

For Mothers and caretakers having under two years children

1. Any mothers and caretakers having under two years children residing in Joshipur Rural Municipality during intervention.

Exclusion Criteria:

Who not available during the time of data collection

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Acceptability of Health Workers Training using key informant interview | At three months
  Acceptability includes the attitude and perception of health workers regarding Health workers training and satisfaction level of health workers attending Health workers training on GMP guidelines. For which, a qualitative method (KII) with health workers using KII guideline will be employed for information collection among the health workers attending the health worker's Training
Appropriateness of Health workers Training using Key informant interview | At three months
  Appropriateness is defined as Health workers training suitable for the cultural, social and economic context of Joshipur rural municipality and alignment of Health workers training to the needs and preferences of the health workers. For which, Key Informant Interview using KII guideline will be employed for information collection
Feasibility of Health workers Training | At three months
  Feasibility includes practicality and ease of attending health workers training and availability of resources. For which information will be collected from health workers through Key Informant Interview using KII guideline.
Fidelity to GMP steps assed through observing HMIS register | At three months
  Fidelity to GMP steps refers to evaluating the extent to which health workers adhere to the steps of GMP. It will be assessed by observing at the nutrition register by health workers as recoded of the steps conducted for growth monitoring and Promotion.
Acceptability of GMP day | At three months
  Acceptability includes the attitude and perception of mothers and caretakers regarding Growth monitoring and Promotion Day . For which, qualitative method (Focus group discussion, FGD using FGD guideline, In-depth Interview, IDI using IDI guideline) will be employed for information collection.
Appropriateness of GMP day | At three months
  Appropriateness includes the alignment of the Growth monitoring and Promotion Day with the needs and preferences of the target population. For which Qualitative method will be employed for information collection.
Feasibility of GMP day to health workers using key informant interview | At three months
  Feasibility includes practicality and ease of implementing GMP day from health workers in the health facility which will be assessed using Key informant interview with health workers using KII guideline.

CONTACTS AND LOCATIONS:
Overall Officials: Amrita Ghimire, MPH, Principal Investigator — Kathmandu University School of Medical Sciences
Locations (1):
- Joshipur rural Municipality, Joshi̇̄pur, Far Western, Nepal

IPD SHARING:
Plan to Share IPD: No